CLINICAL TRIAL: NCT00709436
Title: Randomized, Multiple-center, Double-blind, Placebo-controlled Study of the Safety and Analgesic Efficacy of Repeated Dosing of PMI-150 (Intranasal Ketamine) to Treat Acute Post-operative Pain Following Orthopedic Trauma, Injury, or Surgery.
Brief Title: Safety and Efficacy of Repeated Doses of PMI-150 (Intranasal Ketamine) in Acute Post-operative Pain Following Orthopedic Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KET-017
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Pain, Postoperative
Keywords: orthopedic; ketamine; pain
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): PMI-150 (intranasal ketamine) at time 0 and specified time points thereafter.
  Interventions: Drug: PMI-150 (intranasal ketamine)
- 2 (Placebo Comparator): Placebo at time 0 and specified time points thereafter.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PMI-150 (intranasal ketamine) — PMI-150 (intranasal ketamine) at time 0 and scheduled times thereafter.
  Arms: 1
Drug: Placebo — Placebo (intranasal) at time 0 and scheduled times thereafter.
  Arms: 2

SUMMARY:
The purpose of this research study is to evaluate the safety and analgesic efficacy of PMI-150 (intranasal ketamine) compared to placebo in patients with acute post-operative pain following orthopedic trauma, injury, or surgery.

DETAILED DESCRIPTION:
Patients will be randomly assigned to PMI-150 (intranasal ketamine) or placebo and will receive repeated doses and be assessed for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* patient is scheduled for elective orthopedic surgery or procedure

Exclusion Criteria:

* patient has received an investigational drug or participated in a clinical trial within 30 days or 5 half-lives (whichever is longer) of entering this study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2008-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Measures of pain intensity difference | 0-6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Javelin Pharmaceuticals, Study Director — Javelin Pharmaceuticals
Locations (16):
- United States (16):
  - Jefferson Clinic, Birmingham, Alabama
  - Shoals Clinical Research, Florence, Alabama
  - Helen Keller Hospital, Sheffield, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Vertex Clinical Research, Bakersfield, California
  - California Clinical Research, Davis, California
  - CORE Orthopedic Medical Center, Encinitas, California
  - JDP Medical, Aurora, Colorado
  - Southeastern Center for Clinical Research, Atlanta, Georgia
  - Chesapeake Research Group, Pasadena, Maryland
  - The Ohio State University, Columbus, Ohio
  - Allegehny Pain Management, Altoona, Pennsylvania
  - University Orthopedics, State College, Pennsylvania
  - Comprehensive Pain Specialists, Hendersonville, Tennessee
  - Scott and White Memorial Hospital, Temple, Texas
  - Jean Brown Research, Salt Lake City, Utah